CLINICAL TRIAL: NCT01514071
Title: Animated Picture to Improve Provider Adherence to CT Scan for Head Injury Rule
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospitals and Clinics of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1103-040
Record Dates: First submitted 2012-01-12; First posted 2012-01-20 (Estimated); Last update posted 2013-07-31 (Estimated); Status verified 2013-07

CONDITIONS: Minor Head Injury
Keywords: head injury; CT; emergency; radiation
MeSH Terms: conditions — Craniocerebral Trauma; Emergencies

ARMS (1):
- Pop-up picture (Experimental)
  Interventions: Behavioral: Pop-up picture

INTERVENTIONS:
Behavioral: Pop-up picture — An animated picture depicting the key elements of the PECARN CT scan head injury rules will be explained. The picture will "pop-up" when a provider selects the order set for a CT scan due to head injury. Providers will need to select a box stating the patient either "meets criteria" or "does not meet criteria" in order to close the animated picture window.

SUMMARY:
It is difficult for Pediatric Emergency Department providers to recognize clinically significant head injuries that are likely to require neurosurgical intervention or close monitoring from those that can be safely discharged.

Research Question How do a combination of education and an animated picture depicting the PECARN CT Head Injury rules impact compliance to these rules and reduce unnecessary head CT scans?

Design This is a within subject, repeated measures study design.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting to Children's ED will be included if they:
* Are between 0 and 18 years of age (inclusive)
* Receive a discharge diagnosis of head injury
* Present to the ED within 24 hours of the head injury
* GCS of 14 or greater

Exclusion Criteria:

* Patients will be excluded if they :
* Had a CT scans done in an outside transferring institution
* Have obvious penetrating head injuries
* Had a trivial injury mechanisms such as ground-level falls or walking or running into stationary objects
* Have no signs or symptoms of head trauma other than scalp abrasions and lacerations.
* Have known brain tumors, pre-existing neurological disorders complicating assessment, ventricular shunts, bleeding disorders

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 746 (Estimated)
Dates: Start 2012-02; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Compliance to the PECARN CT Scan Head Injury rules | 3 months

SECONDARY OUTCOMES:
Decreased rate of CT scans | 3 months

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Children's Hospitals and Clinics of Minnesota, Minneapolis, Minnesota
  - Children's Hospitals and Clinics of Minnesota, Twin Cities, Minnesota

REFERENCES:
- [Background] Kuppermann N, Holmes JF, Dayan PS, Hoyle JD Jr, Atabaki SM, Holubkov R, Nadel FM, Monroe D, Stanley RM, Borgialli DA, Badawy MK, Schunk JE, Quayle KS, Mahajan P, Lichenstein R, Lillis KA, Tunik MG, Jacobs ES, Callahan JM, Gorelick MH, Glass TF, Lee LK, Bachman MC, Cooper A, Powell EC, Gerardi MJ, Melville KA, Muizelaar JP, Wisner DH, Zuspan SJ, Dean JM, Wootton-Gorges SL; Pediatric Emergency Care Applied Research Network (PECARN). Identification of children at very low risk of clinically-important brain injuries after head trauma: a prospective cohort study. Lancet. 2009 Oct 3;374(9696):1160-70. doi: 10.1016/S0140-6736(09)61558-0. Epub 2009 Sep 14. PMID 19758692